CLINICAL TRIAL: NCT04470635
Title: Thiol/Disulphide Homeostasis and Salivary Vascular Endothelial Growth Factor Levels in Type 1 Diabetic Patients With Gingivitis
Brief Title: Thiol/Disulphide Homeostasis and Vascular Endothelial Growth Factor Levels in Diabetic Children
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Assoc.Prof.Dr, Aydin Adnan Menderes University
Other Study IDs: 2020/114
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Periodontal Diseases
Keywords: type 1 diabetes mellitus
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Type 1 diabetes with gingivitis: Children with type 1 diabetes mellitus and gingivitis
  Interventions: Diagnostic Test: ELISA
- Type 1 diabetes with healthy gingiva: Children with type 1 diabetes mellitus and healthy gingiva
  Interventions: Diagnostic Test: ELISA
- Healthy children with gingivitis: Systemically healthy children with gingivitis
  Interventions: Diagnostic Test: ELISA
- Healthy children and healthy gingiva: Systemically healthy children with healthy gingiva
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Saliva sample collection
  Other Names: Thiol/disulphide measurement; Total thiol, native thiol and disulphide level

SUMMARY:
The aim of this study to evaluate the vascular endothelial growth factor level and thiol/disulphide homeostasis in saliva of diabetic children with gingivitis.

DETAILED DESCRIPTION:
Eighty children (44 with type 1 diabetes mellitus and 44 systemically healthy) will be recruited for the study. The children will be divided into four subgroups based on their periodontal and systemic condition: 1) systemically and periodontally healthy children, 2) systemically healthy children with gingivitis, 3) periodontally healthy children with T1DM, and 4) children with T1DM and gingivitis. The plaque index, gingival index, probing pocket depth, will recorded. The vascular endothelial growth factor level determined by ELISA. Native thiol, total thiol and disulphide levels will be measured in saliva.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as type 1 diabetes mellitus
* Age between 7-14 years

Exclusion Criteria:

* Having another systemic problem except type 1 diabetes mellitus
* Children carrying orthodontic appliances

Ages: 7 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Eigthy children will be recuited for the study . The children will be classified into four subgroups based on their periodontal status;
  1) systemically and periodontally healthy children, 2) systemically healthy children with gingivitis (G), 3) periodontally healthy children with T1DM, and 4) children with T1DM and gingivitis . The plaque index, gingival index and probing pocket depth will be recorded. The vascular endothelial growth factor in saliva will be determined by ELISA. Additionally total and native thiao and disulphide levels in saliva will be determined.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Vascular endothelial growth factor level | Baseline
  Vascular endothelial growth factor level in saliva

SECONDARY OUTCOMES:
Thiol/disulphide measurement | Baseline
  Total thiol, native thiol and disulphite level in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Sultan KELES, Assoc.Prof., Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Sultan Keles, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No